CLINICAL TRIAL: NCT06160440
Title: A Phase I, Single-center, Double-blind, Placebo-controlled, Single and Multiple Oral Dose, Tolerability, Pharmacokinetic, and Food Effect Study of SC1011 in Healthy Volunteers
Brief Title: The Safety, Tolerability, and Pharmacokinetic Study of SC1011 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou JOYO Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JYE0101
Record Dates: First submitted 2023-11-04; First posted 2023-12-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Diopathic Pulmonary Fibrosis; Pulmonary Fibrosis
Keywords: Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis; Lung Diseases; Respiratory Tract Diseases
MeSH Terms: conditions — Idiopathic Interstitial Pneumonias; Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A single dose SC1011 50mg（A1） (Experimental): Drug: SC1011 tablet Treatment: No food prior to dosing
  Interventions: Drug: SC1011
- A single dose SC1011 150mg（A2） (Placebo Comparator): Drug: SC1011 tablet Drug: SC1011-matching placebo tablet Treatment: No food prior to dosing
  Interventions: Drug: SC1011
- A single dose SC1011 150 mg（A3） (Experimental): Drug: SC1011 tablet Drug: SC1011-matching placebo tablet Treatment: No food prior to dosing
  Interventions: Drug: SC1011
- A single dose SC1011 300mg（A4） (Experimental): Drug: SC1011 tablet Drug: SC1011-matching placebo tablet Treatment: No food prior to dosing
  Interventions: Drug: SC1011

INTERVENTIONS:
Drug: SC1011 — Each subject in the SAD groups participated in 1 treatment period only and reside at the clinical research unit (CRU) from Day -1 (the day before dosing) to Day 7 (144 hours post dose).

SUMMARY:
The goal of this clinical trial is to learn about the safety, tolerability and pharmacokinetic profiles of SC1011,in health conditions. The main questions it aims to answer are:

Safety and tolerability profiles in healthy subjects.Pharmacokinetic profiles in healthy subjects.Food effect in healthy subjects.Participants will complete the study including screening period, dosing period, and observation period. Researchers will compare the inhibitory activity of SC1011 tablets with pirfenidone capsules against the same biomarkers(e.g. blood TNFα) to see if they are different between the two drugs.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, single, and multiple oral dose study conducted in 2 parts.Part A will comprise a single-dose, sequential-group study incorporating a food effect evaluation. Part B will comprise a multiple-dose, sequential-group study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, of any race, between 18 and 45 years of age, inclusive, at Screening.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive, at Screening.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations at Screening and/or Check-in as assessed by the Investigator.
* Females will be nonpregnant and nonlactating. Females of childbearing potential and male subjects will agree to use contraception.
* Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance.
* Alcohol consumption of > 21 units per week for males and > 14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL wine), or a positive alcohol breath test at Check-in.
* Any screening laboratory or ECG results are not within the normal reference range and are considered clinically significant.
* Participants who participated in other clinical trials within 3 months prior to administration.
* Blood donation or blood loss exceeding 400 mL within 2 months prior to administration.
* Participants who smoked, drank alcohol, tea, food or drink containing xanthine or caffeine, or had strenuous exercise, or had other factors affecting drug absorption, distribution, metabolism and excretion 2 days before drug administration.
* Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and serious adverse events related drug. | Evaluations will be conducted for up to 7 days after first administration
  Adverse events are coded according to the ICH Medical Dictionary of Regulatory Activities (MedDRA 24.0 or above). ADR: Adverse events that are "definitely related, probably related, or undetermined" in relation to the investigational drug.

SECONDARY OUTCOMES:
Geometric Mean of Maximum Observed Plasma Concentration of SC1011 | Evaluations will be conducted for up to 7 days after first administration
  Peak concentration. It was directly obtained from the measured data of blood concentration and time.
Area under the plasma concentration-time curve (AUC) from time zero to infinity of SC1011 | Evaluations will be conducted for up to 7 days after first administration
  The area under the curve extrapolated from zero to infinity. AUC0-∞=AUC0-t+Ct/λz(Ct is the last determinable blood concentration, λz is elimination rate constant).

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guang Zhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No